CLINICAL TRIAL: NCT02551718
Title: Individualized Treatment for Relapsed/Refractory Acute Leukemia Based on Chemosensitivity and Genomics/Gene Expression Data
Brief Title: High Throughput Drug Sensitivity Assay and Genomics- Guided Treatment of Patients With Relapsed or Refractory Acute Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary-Beth Percival, Assistant Professor, Division of Hematology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9226; NCI-2015-01299 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9226 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1015012 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2015-08-25; First posted 2015-09-16 (Estimated); Results first posted 2021-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Recurrent Acute Leukemia of Ambiguous Lineage; Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Lymphoblastic Leukemia; Refractory Acute Myeloid Leukemia; Refractory Acute Leukemia of Ambiguous Lineage
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Gene Expression Profiling; Genetic Variation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemosensitivity testing, chemotherapy) (Experimental): Leukemia cells purified from blood or bone marrow samples are analyzed for sensitivity to individual drugs and drug combination and by next generation sequencing.
  Interventions: Other: Chemosensitivity Assay; Other: Cytology Specimen Collection Procedure; Genetic: Gene Expression Analysis; Genetic: Genetic Variation Analysis; Drug: In Vitro Sensitivity-Directed Chemotherapy

INTERVENTIONS:
Other: Chemosensitivity Assay — Lab test in which leukemia cells obtained from blood or bone marrow are tested for sensitivity to 115 drugs individually and in certain combinations
  Other Names: Chemosensitivity Testing
Other: Cytology Specimen Collection Procedure — Undergo blood or bone marrow collection
  Other Names: Cytologic Sampling
Genetic: Gene Expression Analysis — Analysis of leukemia cell genes to identify possible drug targets
Genetic: Genetic Variation Analysis — Analysis of leukemia cell genes to identify possible drug targets
  Other Names: Genetic Variation; GENVAR; mutation analysis
Drug: In Vitro Sensitivity-Directed Chemotherapy — Receive personalized chemotherapy with one or more of the following drugs:
  Afatinib Arsenic trioxide Axitinib Azacitidine Bexarotene Bortezomib Bosutinib Busulfan Cabazitaxel Cabozantinib Carfilzomib Ceritinib Cladribine Clofarabine Crizotinib Cytarabine HCl Dabrafenib Dasatinib Daunorubicin HCl Decitabine Erlotinib Etoposide Everolimus Fludarabine Gefitinib Gemcitabine HCl Hydroxyurea Imatinib Irinotecan Lapatinib Lomustine Melphalan Mercaptopurine Methotrexate Mitoxantrone Nelarabine Nilotinib Paclitaxel Pazopanib Pentostatin Ponatinib Pralatrexate Rapamycin Regorafenib Romidepsin Ruxolitinib Sorafenib Sunitinib Temsirolimus Thioguanine Topotecan HCl Trametinib Tretinoin

SUMMARY:
This pilot clinical trial studies the feasibility of choosing treatment based on a high throughput ex vivo drug sensitivity assay in combination with mutation analysis for patients with acute leukemia that has returned after a period of improvement (relapsed) or does not respond to treatment (refractory). A high throughput screening assay tests many different drugs individually or in combination that kill leukemia cells in tiny chambers at the same time. High throughput drug sensitivity assay and mutation analysis may help guide the choice most effective for an individual's acute leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test patient cells in a high throughput assay against individual drugs and drug combinations within 21 days to enable optimal choice of drug combinations for therapy.

II. To test gene expression that reveals activation of druggable pathways or mutations in genes that confer susceptibility to specific agents may also be considered in choice of treatment.

SECONDARY OBJECTIVE:

I. To evaluate the response to the chosen therapy.

OUTLINE:

Leukemia cells obtained from blood or bone marrow are analyzed for sensitivity to both individual drugs and drug combinations via high throughput chemotherapy sensitivity assay and next generation sequencing assays. Doctors will then recommend chemotherapy regimens based on the results.

After completion of the chemotherapy regimen, patients are followed up at 2-4 weeks for response, and then every 3 months for 2 years for duration of response and survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute leukemia by World Health Organization (WHO) criteria (e.g.-acute myeloid leukemia, acute lymphoblastic leukemia, acute leukemia of ambiguous origin)
* Either:

  * Relapsed after or refractory to prior treatment with at least two regimens or lines of treatment
  * Prior failure of at least one regimen or line of treatment, with poor cytogenetic or other risk factors, and ineligible for other clinical trials
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 3
* Expectation that we can obtain about 10 million blasts from blood and/or marrow (e.g., circulating blast count of 5,000 or greater or cellular marrow with greater than or equal to 20% blasts)
* Bilirubin =< 1.5 x upper limit of normal (ULN) unless elevation is thought to be due to Gilbert's syndrome, hemolysis, or hepatic infiltration by the hematologic malignancy
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SPGT) (alanine aminotransferase [ALT]) =< 2.5 x ULN, unless elevation is thought to be due to hepatic infiltration by the hematologic malignancy
* Alkaline phosphatase =< 2.5 x ULN, unless elevation is thought to be due to hepatic infiltration by the hematologic malignancy
* Serum creatinine =< 2.0 mg/dL
* Informed consent
* Willing to use contraception when appropriate
* Expected survival is greater than 100 days

Exclusion Criteria:

* No other active cancer that requires systemic chemotherapy or radiation
* Active systemic fungal, bacterial, viral or other infection, unless disease is under treatment with antimicrobials and considered controlled in the opinion of the investigator
* Significant organ compromise that will increase risk of toxicity or mortality
* Pregnancy or lactation

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2021-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Elizabeth Percival, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemosensitivity Testing: Leukemia cells purified from blood or bone marrow samples are analyzed for sensitivity to individual drugs and drug combination and by next generation sequencing.
  Chemosensitivity Assay: Lab test in which leukemia cells obtained from blood or bone marrow are tested for sensitivity to 115 drugs individually and in certain combinations
  Cytology Specimen Collection Procedure: Undergo blood or bone marrow collection
  Gene Expression Analysis: Analysis of leukemia cell genes to identify possible drug targets
  Genetic Variation Analysis: Analysis of leukemia cell genes to identify possible drug targets
  In Vitro Sensitivity-Directed Chemotherapy: Receive personalized chemotherapy with one or more of the following drugs:
  Afatinib Arsenic trioxide Axitinib Azacitidine Bexarotene Bortezomib Bosutinib Busulfan Cabazitaxel Cabozantinib Carfilzomib Ceritinib Cladribine Clofarabine Crizotinib Cytarabine HCl Dabrafenib Dasatinib Daunorubicin HCl Decitabine Erlotinib Etoposide Everolimus Fludarabine Gefitinib Gemcitabine HCl Hydroxyurea Imatinib Irinotecan Lapatinib Lomustine Melphalan Mercaptopurine Methotrexate Mitoxantrone Nelarabine Nilotinib Paclitaxel Pazopanib Pentostatin Ponatinib Pralatrexate Rapamycin Regorafenib Romidepsin Ruxolitinib Sorafenib Sunitinib Temsirolimus Thioguanine Topotecan HCl Trametinib Tretinoin
Period: Overall Study
Arm/Group | Chemosensitivity Testing
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemosensitivity Testing
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 11
Age, Continuous [Mean (Full Range); unit: years] | 54 [23 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients we Are Able to Test and Initiate Treatment Within a 21 Day Period
Description: The study will be considered successful (feasibility demonstrated) if it is possible to choose and initiate a combination drug regimen within 21 days in 9 out of 15 patients. With that outcome, there would be 90% confidence that the true feasibility rate is at least 40%.
Time Frame: Up to 21 days
Measure: Count of Participants; unit: Participants
Groups:
- Chemosensitivity Testing and Treatment Initiation Within 21 Days: Leukemia cells purified from blood or bone marrow samples are analyzed for sensitivity to individual drugs and drug combination and by next generation sequencing.
  Chemosensitivity Assay: Lab test in which leukemia cells obtained from blood or bone marrow are tested for sensitivity to 115 drugs individually and in certain combinations
  Cytology Specimen Collection Procedure: Undergo blood or bone marrow collection
  Gene Expression Analysis: Analysis of leukemia cell genes to identify possible drug targets
  Genetic Variation Analysis: Analysis of leukemia cell genes to identify possible drug targets
  In Vitro Sensitivity-Directed Chemotherapy: Receive personalized chemotherapy with one or more of the following drugs:
  Afatinib Arsenic trioxide Axitinib Azacitidine Bexarotene Bortezomib Bosutinib Busulfan Cabazitaxel Cabozantinib Carfilzomib Ceritinib Cladribine Clofarabine Crizotinib Cytarabine HCl Dabrafenib Dasatinib Daunorubicin HCl Decitabine Erlotinib Etoposide Everolimus Fludarabine Gefitinib Gemcitabine HCl Hydroxyurea Imatinib Irinotecan Lapatinib Lomustine Melphalan Mercaptopurine Methotrexate Mitoxantrone Nelarabine Nilotinib Paclitaxel Pazopanib Pentostatin Ponatinib Pralatrexate Rapamycin Regorafenib Romidepsin Ruxolitinib Sorafenib Sunitinib Temsirolimus Thioguanine Topotecan HCl Trametinib Tretinoin
Arm/Group | Chemosensitivity Testing and Treatment Initiation Within 21 Days
Number analyzed (Participants) | 34
Participants | 21

2. Secondary Outcome: Rate of Complete Remission
Description: The secondary objective is to evaluate the response to the chosen therapy. Response will be evaluated using European LeukemiaNet Response Evaluation Criteria in AML (2010 version)
Time Frame: Up to 2 years
Population: Number of complete remissions + complete remissions with incomplete blood counts
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Chemosensitivity Testing, Chemotherapy): Leukemia cells purified from blood or bone marrow samples are analyzed for sensitivity to individual drugs and drug combination and by next generation sequencing.
  Chemosensitivity Assay: Lab test in which leukemia cells obtained from blood or bone marrow are tested for sensitivity to 115 drugs individually and in certain combinations
  Cytology Specimen Collection Procedure: Undergo blood or bone marrow collection
  Gene Expression Analysis: Analysis of leukemia cell genes to identify possible drug targets
  Genetic Variation Analysis: Analysis of leukemia cell genes to identify possible drug targets
  In Vitro Sensitivity-Directed Chemotherapy: Receive personalized chemotherapy with one or more of the following drugs:
  Afatinib Arsenic trioxide Axitinib Azacitidine Bexarotene Bortezomib Bosutinib Busulfan Cabazitaxel Cabozantinib Carfilzomib Ceritinib Cladribine Clofarabine Crizotinib Cytarabine HCl Dabrafenib Dasatinib Daunorubicin HCl Decitabine Erlotinib Etoposide Everolimus Fludarabine Gefitinib Gemcitabine HCl Hydroxyurea Imatinib Irinotecan Lapatinib Lomustine Melphalan Mercaptopurine Methotrexate Mitoxantrone Nelarabine Nilotinib Paclitaxel Pazopanib Pentostatin Ponatinib Pralatrexate Rapamycin Regorafenib Romidepsin Ruxolitinib Sorafenib Sunitinib Temsirolimus Thioguanine Topotecan HCl Trametinib Tretinoin
Arm/Group | Treatment (Chemosensitivity Testing, Chemotherapy)
Number analyzed (Participants) | 34
Participants | 5

3. Secondary Outcome: Survival
Description: Disease free and overall survival data will be assessed by contacting the referring MD or the patient every three months for the first two years.
Time Frame: Up to 2 years
Population: Overall survival in months from date of study consent
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Treatment (Chemosensitivity Testing, Chemotherapy)
Number analyzed (Participants) | 34
months | 6.91 (7.64)

ADVERSE EVENTS:
Time Frame: 5 years
Description: Non-hematologic toxicities >/= grade 3 were recorded from time of assay-guided therapy administration through 14 days after last administration of study therapy Hospitalizations or prolongation of hospitalizations for protocol-scheduled procedures, blood product transfusions, or for social reasons (i.e. awaiting transport home) were not considered SAEs. And hospitalization or prolongation of hospitalizations for fever and/or infection were considered expected, and not considered SAEs.
Arm/Group | Chemosensitivity Testing
All-Cause Mortality (participants affected / at risk) | 32/34
Serious Adverse Events (participants affected / at risk) | 11/34
Other Adverse Events (participants affected / at risk) | 26/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemosensitivity Testing (N=34)
Anaphylaxis (Immune system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Enterobacter Cloacae Sepsis (Infections and infestations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypoxemic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Neutropenic fever with Sepsis Physiology (Infections and infestations) | 1 (1)
Intermittent Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Pneumonia (Infections and infestations) | 2 (2)
Pain (General disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhizopus Pneumonia (Infections and infestations) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemosensitivity Testing (N=34)
Atrial Fibrillation with RVR (Cardiac disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (2)
Anorectal Infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Bacteremia Infection (Infections and infestations) | 1 (1)
C. Diff Colitis with Diarrhea (Gastrointestinal disorders) | 1 (2)
Catheter Related Infection (Infections and infestations) | 1 (1)
Central Line Associated DVT (Vascular disorders) | 1 (1)
Coag Negative Staph Bacteremia (Infections and infestations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Distributive Shock (Infections and infestations) | 1 (1)
Enterocolitis (Infections and infestations) | 2 (2)
Eye Infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 10 (19)
Granulicatella Adiacens Bacteremia (Infections and infestations) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Hyperbilirubinemia (Investigations) | 2 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4)
INR Increased (Investigations) | 1 (1)
Invasive Fungal Sinusitis (Infections and infestations) | 1 (1)
Lung Infection (Infections and infestations) | 3 (3)
Oral Mucositis (Infections and infestations) | 2 (2)
Pain (General disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pseudomonas Bacteremia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 1 (1)
Rothia Mucilaginosa Bacteremia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (4)
Staph Epidermidis Bacteremia (Infections and infestations) | 2 (2)
Staphylococcus Infection (Infections and infestations) | 1 (1)
Stenotrophomonas Maltophilia Bacteremia (Infections and infestations) | 1 (1)
Subdural Hematoma (Blood and lymphatic system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transaminitis (Investigations) | 1 (1)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT02551718/Prot_SAP_000.pdf